CLINICAL TRIAL: NCT06131905
Title: Magnesium Sulfate as an Adjuvant to Propofol During Consious Sedation in Adult Patients Undergoing Colonoscopy
Brief Title: Magnesium Sulfate as an Adjuvant to Propofol During Consious Sedation in Colonoscopy
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Sayed Mahmoud Sayed, Doctor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Magnesium in colonoscopy
Record Dates: First submitted 2023-11-02; First posted 2023-11-14 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Magnesium; Intraoperative Analgesia
MeSH Terms: interventions — Magnesium Sulfate; Propofol

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group M (Magnesium sulfate+Propofol) (Active Comparator): Includes thirdy patients receive 40mg /kg magnesium sulfate diluted with normal saline to a total volume of 100 ml plus ,An initial bolus dose of 1 mg/kg propofol was administered over 30 is followed by a continuous intravenous infusion of propofol at a maintenance dose of 2 mg/kg/h
  Interventions: Drug: Magnesium Sulfate; Drug: Propofol
- Group N (Propofol) (Active Comparator): Includes thirdy patients receive an equal volume of normal saline as a placebo.plus An initial bolus dose of 1 mg/kg propofol was administered over 30 is followed by a continuous intravenous infusion of propofol at a maintenance dose of 2 mg/kg/h
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Magnesium Sulfate — 40 mg/kg magnesium sulfate diluted with normal saline to a total volume of 100 ml was administered for 15 min.plus ,An initial bolus dose of 1 mg/kg propofol was administered over 30 is followed by a continuous intravenous infusion of propofol at a maintenance dose of 2 mg/kg/h
  Arms: Group M (Magnesium sulfate+Propofol)
Drug: Propofol — An initial bolus dose of 1 mg/kg propofol was administered over 30 is followed by a continuous intravenous infusion of propofol at a maintenance dose of 2 mg/kg/h

SUMMARY:
Colonoscopy is one of the most commonly performed outpatient procedures throughout the world as a screening, diagnostic, and therapeutic tool to evaluate the large intestine from the distal rectum to the cecum.Propofol is the most commonly used hypnotic agent in sedation during endoscopic procedures for its advantages of fast onset and quick recovery. However, propofol may cause respiratory depression and cardiovascular events, which are easier to appear in cases of old age and high speed administration of propofol.Magnesium is a non-specific calcium channel inhibitor and a non-competitive N-methyl-D-aspartate(NMDA)receptor antagonist, which has analgesic and mild sedative properties .

DETAILED DESCRIPTION:
Colonoscopy is one of the most commonly performed outpatient procedures throughout the world as a screening, diagnostic, and therapeutic tool to evaluate the large intestine from the distal rectum to the cecum . Colonoscopy is currently an important examination method for colorectal diseases. It can provide clear images of lesions and provide biopsy for biopsy. It can improve the accuracy and sensitivity of colorectal cancer diagnosis .The most common complications in gastrointestinal endoscopy are not related to the procedure, but they are related to sedation; they include cardio- respiratory adverse events such as hypoxemia, hypoventilation, apnea, dysrhythmias, hypotension and vasovagal episodes .Propofol is the most commonly used hypnotic agent in sedation during endoscopic procedures for its advantages of fast onset and quick recovery. However, propofol may cause respiratory depression and cardiovascular events, which are easier to appear in cases of old age and high speed administration of propofol . Moreover, high doses of propofol may cause dose-dependent hemodynamic instability in older or feeble patients. Therefore, it is essential to minimize the dosage of propofol to prevent cardiopulmonary complications associated with sedation, especially in the elderly, by combining with an adjuvant medication. Although benzodiazepines or opioids combined with propofol can reduce the consumption of propofol, elderly patients usually feature a higher overall body fat content than younger patients which may delay the metabolism of lipid-soluble propofol, opioid, and benzodiazepines . Magnesium is the fourth most plentiful cation in the body and the second most plentiful intracellular cation after potassium. Approximately one half of total body magnesium is present in bone and 20% in skeletal muscle. Magnesium is necessary for the presynaptic release of acetylcholine from nerve endings and may produce effects similar to calcium-entry-blocking drugs . Magnesium is a non-specific calcium channel inhibitor and a non-competitive N-methyl-D-aspartate(NMDA)receptor antagonist, which has analgesic and mild sedative properties . It has been demonstrated that intravenous administration of magnesium sulfate can reduce the overall use of intraoperative propofol and the postoperative analgesia requirement effectively in various types of surgery .These findings implied that magnesium sulfate may be used as a promising adjuvant drug for colonoscopy sedation due to its analgesic and sedative properties .

ELIGIBILITY:
Inclusion Criteria:

* 1. The subject is scheduled for elective colonoscopy. 2. The subject is ≥ 40 years and ≤ 70 years. 3. Both sexes. 4.No obvious abnormalities in preoperative ECG, blood routine, electrolytes, and other tests. 5. ASA class 1-3.

Exclusion Criteria:

* 1.Subject is known or believed to be pregnant or lactating women. 2. Patients are known hypersensitivity to any of the drugs that would be used in the study. 3. Severe cardiac, renal, lung, or liver diseases. 4. Hypotension (systolic blood pressure< 90 mm Hg), uncontrolled hypertension (systolic blood pressure> 170 mmHg, diastolic blood pressure> 100mmHg). 5. Chronic Opioid Use (daily or almost daily use of opioids for> 3 months). 6. Patients that are immunologically compromised. 7. Sleep apnea syndrome or difficult airway. 8. preexisting hypoxemia (Spo2< 90 %). 9. History of adverse events with prior sedation. Additionally, patients who had taken any sedative drugs within the previous 24h

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Total consumption of propfol | During procedure
  Calculate the total dose of propofol used for each case

SECONDARY OUTCOMES:
sedation time | During procedure and One hour after procedure
  Measure sedation time during and after procedure

CONTACTS AND LOCATIONS:
Overall Officials: Essam Mohamed Manna, Professor, Study Chair — Professor of Anesthesia and Intensive Care, Faculty of Medicine, Assiut University; Raja Ahmad Abdullah Mohamed, Study Director — Assistant Professor of Anesthesia and Intensive Care, Faculty of Medicine, Assiut University

REFERENCES:
- [Background] Liu J, Liu X, Peng LP, Ji R, Liu C, Li YQ. Efficacy and safety of intravenous lidocaine in propofol-based sedation for ERCP procedures: a prospective, randomized, double-blinded, controlled trial. Gastrointest Endosc. 2020 Aug;92(2):293-300. doi: 10.1016/j.gie.2020.02.050. Epub 2020 Mar 7. PMID 32156544
- [Background] Lu Z, Li W, Chen H, Qian Y. Efficacy of a Dexmedetomidine-Remifentanil Combination Compared with a Midazolam-Remifentanil Combination for Conscious Sedation During Therapeutic Endoscopic Retrograde Cholangio-Pancreatography: A Prospective, Randomized, Single-Blinded Preliminary Trial. Dig Dis Sci. 2018 Jun;63(6):1633-1640. doi: 10.1007/s10620-018-5034-3. Epub 2018 Mar 29. PMID 29594976
- [Background] Herroeder S, Schonherr ME, De Hert SG, Hollmann MW. Magnesium--essentials for anesthesiologists. Anesthesiology. 2011 Apr;114(4):971-93. doi: 10.1097/ALN.0b013e318210483d. PMID 21364460
- [Background] Olgun B, Oguz G, Kaya M, Savli S, Eskicirak HE, Guney I, Kadiogullari N. The effects of magnesium sulphate on desflurane requirement, early recovery and postoperative analgesia in laparascopic cholecystectomy. Magnes Res. 2012 Jul;25(2):72-8. doi: 10.1684/mrh.2012.0315. PMID 22728648
- [Background] De Oliveira GS, Bialek J, Fitzgerald P, Kim JY, McCarthy RJ. Systemic magnesium to improve quality of post-surgical recovery in outpatient segmental mastectomy: a randomized, double-blind, placebo-controlled trial. Magnes Res. 2013 Oct-Dec;26(4):156-64. doi: 10.1684/mrh.2014.0349. PMID 24491463
- [Result] Rex DK, Khalfan HK. Sedation and the technical performance of colonoscopy. Gastrointest Endosc Clin N Am. 2005 Oct;15(4):661-72. doi: 10.1016/j.giec.2005.08.003. PMID 16278131
- [Result] Wernli KJ, Brenner AT, Rutter CM, Inadomi JM. Risks Associated With Anesthesia Services During Colonoscopy. Gastroenterology. 2016 Apr;150(4):888-94; quiz e18. doi: 10.1053/j.gastro.2015.12.018. Epub 2015 Dec 18. PMID 26709032
- [Result] Cote GA, Hovis RM, Ansstas MA, Waldbaum L, Azar RR, Early DS, Edmundowicz SA, Mullady DK, Jonnalagadda SS. Incidence of sedation-related complications with propofol use during advanced endoscopic procedures. Clin Gastroenterol Hepatol. 2010 Feb;8(2):137-42. doi: 10.1016/j.cgh.2009.07.008. Epub 2009 Jul 14. PMID 19607937